CLINICAL TRIAL: NCT00042042
Title: Screening Adolescents for Type 2 Diabetes Mellitus in a Community Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Duke University (Other); Diabetes Trust Fund (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: NCRR-M01RR00030-0199
Record Dates: First submitted 2002-07-22; First posted 2002-07-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Behavioral: Family based educational program

SUMMARY:
The purpose of this study is to evaluate the prevalence of Type 2 diabetes or impaired glucose tolerance in a subset of children 10-19 years of age in an inner city community clinic. The demographics of the clinic are 75% African American, 20% Hispanic, 5% other. African American and Hispanic patients have a higher prevalence of diabetes with significant morbidity, predominantly from microvascular and macrovascular disease. Obesity is commonly seen in patients with Type 2 diabetes and contributes to the underlying insulin resistance seen in the disease. Obesity is an increasing health problem among adolescents. Since Type 2 diabetes can be present for several years before diagnosis, it is worrisome that younger children will have undiagnosed Type 2 diabetes for years. This will increase the risk of earlier complications in these patients as young adults.

We hypothesize that the occurrence of abnormal glucose metabolism in 400 children with either a history of obesity, family history of diabetes mellitus, or symptoms suggestive of diabetes mellitus will be higher than the general pediatric population. We believe that a family based educational program can reduce fasting plasma glucose.

DETAILED DESCRIPTION:
This is a two part study. The first part is a diabetes screening study of 400 adolescent children who have a risk factor for type 2 diabetes to determine the prevalence of abnormal glucose metabolism in such patients. At the time of glucose screening all children will be given a dietary habit survey and two measures of depression/self-esteem to complete so that we may measure the correlation of depression and obesity and depression and abnormal glucose metabolism.

The second part tests the efficacy of a family based educational program in lowering fasting glucose in children who screen positive for type 2 DM, hyperinsulinemia, or impaired glucose tolerance. This educational assessment will be administered in an observational non-randomized, non-blinded fashion. The dietary habit survey and the measures of self-esteem and depression will aid us in creating this family based educational study.

ELIGIBILITY:
Inclusion criteria for screening will be patients who have one of the following:

1. 120% of ideal body weight or BMI> 27
2. Weight greater than 75th percentile
3. Family history of type 2 diabetes in first or second degree relative
4. Acanthosis nigricans or skin tags as signs of insulin resistance
5. Symptoms of hyperglycemia (polyuria, polydipsia, polyphagia, or recurrent infections).
6. Symptoms or signs of PCOS (hyperandrogenism, hirsutism, irregular menses)

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States